CLINICAL TRIAL: NCT02129647
Title: Phase II Study of Axitinib in Patients With Neurofibromatosis Type 2 and Progressive Vestibular Schwannomas
Brief Title: Study of Axitinib in Patients With Neurofibromatosis Type 2 and Progressive Vestibular Schwannomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-00004
Record Dates: First submitted 2014-04-29; First posted 2014-05-02 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Neurofibromatosis Type 2; Vestibular Schwannomas
Keywords: Neurofibromatosis Type 2; Vestibular Schwannomas; Axitinib
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axitinib (Experimental): 5 mg axitinib orally twice daily, with increase to 7 mg orally twice daily and 10 mg orally twice daily after 2 and 4 weeks, respectively, provided no adverse reactions (i.e., not exceeding grade 2 toxicities) and normotensive and not receiving antihypertension medications. Axitinib will be given continuously in 28-day cycles until disease progression or unacceptable toxicity.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib
  Other Names: Inlyta

SUMMARY:
The purpose of this study is to determine if the study drug, AXITINIB, has any effect on tumors found in patients with Neurofibromatosis Type 2 (NF2).

DETAILED DESCRIPTION:
NF2 is a condition that mainly affects the skin and nervous system. It causes non-cancerous tumors to grow on the nerves around a person's body. Some signs of NF2 include a gradual loss of hearing and tumors growing on the skin, the brain and the spinal cord, which can lead to complications.

AXITINIB is an oral drug (taken by mouth) that is approved by the United States Food and Drug Administration (FDA) for the treatment of other types of tumors. However, in this research study, AXITINIB is considered investigational because it is not approved by the FDA for treatment of NF2. Much is known regarding how well it is tolerated (handled), but investigators do not know if it is effective in treating NF2.

This research study will test whether AXITINIB may shrink tumors commonly found in patients with NF2 or stop them from growing. This will help to decide if AXITINIB should be used to treat NF2 patients in the future. AXITINIB is a drug that has been used to treat various forms of cancer. It has not been studied for the treatment of tumors in NF2 patients. Investigators have selected AXITINIB for this clinical trial in patients with NF2 and NF2-related tumors because a very similar drug, bevacizumab, can shrink Vestibular Schwannomas (VS) in some NF2 patients.

Pfizer, Inc., the manufacturer of the study drug, AXITINIB, will provide the AXITINIB being used in this study.

Primary Objective: To estimate the objective volumetric response rates to axitinib in adult NF2 patients with VS.

Secondary Objectives: To assess the toxicity of axitinib given daily in patients with NF2 and to examine the association of objective measures of response on MRI, i.e. volumetric tumor analysis with clinical measures of response, i.e. (audiogram), as well as quality of life assessments (NFTI-QOL). In addition, response in non-VS tumors, such as other schwannomas and meningiomas, may be explored.

ELIGIBILITY:
Inclusion criteria

* Age ≥18 years
* Meets clinical diagnostic criteria for NF2
* At least one volumetrically measurable and ≥1 cc NF2-related VS (histological confirmation not required)
* MRI evidence of progression (either as >2 mm increase in maximum linear diameter on conventional MRI, or a >20%volume increase by 3D volumetrics) over the past ≤18 months, OR progressive hearing loss, defined as a decline in word recognition score below the 95% critical difference interval from baseline score related to VS (i.e., not due to prior interventions such as surgery or radiation)
* Karnofsky performance status (PS) 60-100%. Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Adequate bone marrow function as shown by: absolute neutrophil count ≥1.5 x 10^9/L, Platelets ≥100 x 10^9/L, Hb >9 g/dL
* Adequate liver function as shown by:
* serum bilirubin ≤1.5 x upper limit of normal (ULN)
* ALT and AST ≤2.5x ULN
* INR ≤1.5. (anticoagulation with low molecular weight heparin is allowed if on a stable dose for >2 weeks at time of enrollment.)
* Adequate renal function: serum creatinine ≤1.5 x ULN
* Fully recovered from acute toxic effects of any prior chemotherapy, biological modifiers or radiotherapy
* Any neurologic deficits must be stable for ≥1 week
* Able to provide signed informed consent Exclusion criteria
* Patients currently receiving medical anticancer therapies or who have received medical anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, antibody based therapy, etc.)
* Radiation therapy to a study target tumor within 1 year prior to enrollment, or any radiation therapy within 4 weeks prior to enrollment.
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with bevacizumab or other agents targeting vascular endothelial growth factor (VEGF) or VEGF receptor
* Prior treatment with any investigational drug within the preceding 4 weeks
* Unstable or rapidly progressive disease, including patients who require glucocorticoids for symptomatic control of brain or spinal tumors
* Treatment with strong CYP3A4 enzyme inhibitors or inducers, including but not limited to ketoconazole, itraconazole, ritonavir, phenytoin, carbamazepine, rifampin, rifabutin, phenobarbital and St. John's wort
* Requirement of therapeutic anticoagulant therapy with oral vitamin K antagonists; low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed; therapeutic use of low molecular weight heparin (or similar parenteral drug) for venous-thromboembolic disease is allowed.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Symptomatic congestive heart failure of New York heart Association Class III or IV
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* severely impaired lung function as defined as spirometry and diffusion capacity of lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or O2 saturation that is 90% or less at rest on room air
* active (acute or chronic) or uncontrolled severe infections
* liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of axitinib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes. (Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to administration of axitinib)
* Male patient whose sexual partner(s) are women of child bearing potential, who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Nicolaides, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: 5 mg axitinib orally twice daily, with increase to 7 mg orally twice daily and 10 mg orally twice daily after 2 and 4 weeks. Axitinib will be given continuously in 28-day cycles until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Axitinib
Started | 13
Completed | 10
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — surgical intervention for clinically progressive disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 39 [21 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Expression Levels of p-S6 Based Immunohistochemistry (Histoscore)
Description: The histoscore is given as the sum of the percentage of staining multiplied by an ordinal value corresponding to the intensity level (0 = none, 1 = weak, 2 = moderate, 3 = strong). With 4 intensity levels, the resulting score ranged from 0 (no staining in the tumor) to 300 (diffuse intense staining of the tumor).
Time Frame: 10 days
Measure: Median (Full Range); unit: score
Arm/Group | Axitinib
Number analyzed (Participants) | 10
score | 90 [0 to 220]
Statistical Analysis 1: Comparison: Axitinib; Test type: Other; 10 tissue matched historical controls were analyzed. The Median (Full Range) of the histoscore was 122 (60 to 265)

2. Primary Outcome: Expression Levels of p-ERK Based Immunohistochemistry (Histoscore)
Description: as for outcome 1
Time Frame: 10 days
Measure: Median (Full Range); unit: score
Arm/Group | Axitinib
Number analyzed (Participants) | 10
score | 180 [40 to 220]
Statistical Analysis 1: Comparison: Axitinib; Test type: Other; 10 tissue matched historical controls were analyzed. The Median (Full Range) of the histoscore was 135 (100 to 240)

3. Primary Outcome: Expression Levels of p-AKT Based Immunohistochemistry (Histoscore)
Description: as for outcome 1
Time Frame: 10 days
Measure: Median (Full Range); unit: score
Arm/Group | Axitinib
Number analyzed (Participants) | 10
score | 42 [5 to 100]
Statistical Analysis 1: Comparison: Axitinib; Test type: Other; 10 tissue matched historical controls were analyzed. The Median (Full Range) of the histoscore was 12 (0 to 100)

4. Primary Outcome: Pre-Operative Everolimus Blood Levels
Time Frame: Baseline
Population: No controls - Given that only a single surgery is generally performed to resect meningiomas and schwannomas without prior biopsy, obtaining matched control of pre and post treatment samples from the same tumor was not feasible. The study team therefore relied on matched archival control tissue for comparisons of other outcome measures; Everolimus blood levels not being one of them.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Axitinib
Number analyzed (Participants) | 10
ng/ml | 17.4 [6.9 to 49.6]

5. Primary Outcome: Post-Operative Everolimus Blood Levels
Time Frame: 10 days
Population: as for outcome 4
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Axitinib
Number analyzed (Participants) | 10
ng/ml | 9.4 [6.3 to 43.4]

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Axitinib
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (N=10)
Mucositis (Gastrointestinal disorders) | 3 (3)
nausea (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT02129647/Prot_SAP_000.pdf